CLINICAL TRIAL: NCT04387890
Title: Serologic Surveillance for SARS-CoV-2 (COVID-19) in a Prospective Cohort of Health Care
Brief Title: Serologic Surveillance for SARS-CoV-2 (COVID-19) in a Prospective Cohort of Health Care Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Diego Hernan Giunta, PhD, MPH, MD, MD, MPH, University SoTL, PhD, Hospital Italiano de Buenos Aires
Other Study IDs: 5566
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; SARS-CoV 2; Health Personnel
Keywords: SARS Virus; SARS-CoV-2; COVID-19; Health Personnel
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Serologic Screening: Participants will be screened for IgM and IgG SARS-CoV-2 antibodies at baseline and every 2 weeks. Participants showing symptoms compatible with COVID-19 will undergo nasopharyngeal swab for PCR testing for diagnosis. Participants recovered from COVID-19 will have to have 2 negative and consecutive nasopharyngeal swab PCR tests in order to return to work.
  Interventions: Diagnostic Test: Serologic SARS-CoV-2 screening

INTERVENTIONS:
Diagnostic Test: Serologic SARS-CoV-2 screening — Quantitative Indirect Chemiluminescence Immunoassay (CLIA) to access SARS-CoV-2 specific IgM and IgG serum antibody level every 2 weeks during follow up

SUMMARY:
The investigators will follow a single prospective cohort of 50 Health Care Workers in the Hospital Italiano de Buenos Aires (Argentina) from May 15th to August 31st 2020 using antibody testing for SARS-CoV-2 IgM and IgG at baseline and every 2 weeks in order to assess the incidence of COVID-19, the prevalence of anti-SARS-CoV-2 antibodies (IgM and IgG) and incidence of reinfection or reactivations of previous COVID-19 using viral gene sequencing in this cohort.

DETAILED DESCRIPTION:
SARS-CoV-2 infection in healthcare workers (HCW) is nowadays a frequent problem for patient care and organization of care teams. SARS-CoV-2 antibody assessment provides a tool to evaluate antibody prevalence in hospital staff identifying previously exposed individuals. Serologic testing could identify new cases of COVID-19 in an early fashion and could help to investigate cases of reactivation or reinfection in hospital workers. The study purpose is to conduct a study using serological screening for health care workers in a University Hospital in Buenos Aires in order to assess the risk of COVID-19 on those who have not developed an immune response against the virus, or to detect it in an early fashion (either pre-symptomatic or asymptomatic). If a study participant is suspected to have potential reinfection or reactivation of COVID-19, the investigators will conduct genome sequencing in order to be able to differentiate each case. The investigators will include 50 participants chosen at random among health care workers from the hospital Emergency Department (ED), Internal Medicine wards, or Critical Care Units who are exposed to COVID-19. Participants who agree to join the study and sign the informed consent form will be screened at baseline for SARS-CoV-2 IgM and IgG antibodies, along with a physical exam and basic laboratory determinations. They will be re-screened with antibodies every 2 weeks for a total of 3 months. If they contract COVID-19, antibody determinations and nasopharyngeal swabs will be carried out in order to identify those who are in favorable conditions to return to work. The main objective is to prospectively determine the incidence of COVID-19, Anti SARS-CoV-2 antibody prevalence, and incidence of SARS-CoV-2 reinfection or reactivation of COVID-19 in a health care workers cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare staff (Physicians) AND
2. Directly involved in care of patients with confirmed or suspected COVID-19 AND
3. Working in any of the two hospital venues (Hospital Italiano Central and Hospital Italiano San Justo Agustín Rocca).

Exclusion Criteria:

1. Refusal to sign the Informed Consent Form OR
2. Experienced symptoms compatible with COVID-19 in the last 14 days prior to eligibility screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians directed involved with the healthcare of COVID-19 patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anti SARS-CoV-2 antibodies (IgM and IgG) in health personnel | Baseline at study inclussion
  Patients that has a positive result for IgM or IgG at baseline first test
COVID-19 incidence through serology-based screening and/or compatible symptoms in health personnel previously known to be unexposed to the virus | During 3 months follow up
  Patients that has a positive result for IgM or IgG or PCR during follow up
Incidence of reactivation/reinfection for COVID-19 in health personnel with a positive serology for SARS-CoV-2 | During 3 months follow up
  Patients with confirmed previous SARS Cov 2 antibodies that reactivate symptomons or new increase in antibodies title during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Peroni, MD, Principal Investigator — HIBA; Vanina Stanek, MD, Principal Investigator — HIBA; Diego Sanchez Thomas, MD, Principal Investigator — HIBA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] The Lancet. COVID-19: protecting health-care workers. Lancet. 2020 Mar 21;395(10228):922. doi: 10.1016/S0140-6736(20)30644-9. No abstract available. PMID 32199474
- [Result] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Result] Kimball A, Hatfield KM, Arons M, James A, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Chisty Z, Bell JM, Methner M, Harney J, Jacobs JR, Carlson CM, McLaughlin HP, Stone N, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Russell D, Hiatt B, Gant J, Duchin JS, Clark TA, Honein MA, Reddy SC, Jernigan JA; Public Health - Seattle & King County; CDC COVID-19 Investigation Team. Asymptomatic and Presymptomatic SARS-CoV-2 Infections in Residents of a Long-Term Care Skilled Nursing Facility - King County, Washington, March 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):377-381. doi: 10.15585/mmwr.mm6913e1. PMID 32240128
- [Result] Chu DKW, Pan Y, Cheng SMS, Hui KPY, Krishnan P, Liu Y, Ng DYM, Wan CKC, Yang P, Wang Q, Peiris M, Poon LLM. Molecular Diagnosis of a Novel Coronavirus (2019-nCoV) Causing an Outbreak of Pneumonia. Clin Chem. 2020 Apr 1;66(4):549-555. doi: 10.1093/clinchem/hvaa029. PMID 32031583
- [Result] Yu F, Yan L, Wang N, Yang S, Wang L, Tang Y, Gao G, Wang S, Ma C, Xie R, Wang F, Tan C, Zhu L, Guo Y, Zhang F. Quantitative Detection and Viral Load Analysis of SARS-CoV-2 in Infected Patients. Clin Infect Dis. 2020 Jul 28;71(15):793-798. doi: 10.1093/cid/ciaa345. PMID 32221523
- [Result] Yuan J, Kou S, Liang Y, Zeng J, Pan Y, Liu L. Polymerase Chain Reaction Assays Reverted to Positive in 25 Discharged Patients With COVID-19. Clin Infect Dis. 2020 Nov 19;71(16):2230-2232. doi: 10.1093/cid/ciaa398. PMID 32266381
- [Result] Li Y, Yao L, Li J, Chen L, Song Y, Cai Z, Yang C. Stability issues of RT-PCR testing of SARS-CoV-2 for hospitalized patients clinically diagnosed with COVID-19. J Med Virol. 2020 Jul;92(7):903-908. doi: 10.1002/jmv.25786. Epub 2020 Apr 5. PMID 32219885
- [Result] Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill. 2020 Mar;25(10):2000180. doi: 10.2807/1560-7917.ES.2020.25.10.2000180. PMID 32183930
- [Result] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Result] Elbe S, Buckland-Merrett G. Data, disease and diplomacy: GISAID's innovative contribution to global health. Glob Chall. 2017 Jan 10;1(1):33-46. doi: 10.1002/gch2.1018. eCollection 2017 Jan. PMID 31565258
- [Result] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Result] Hu Z, Song C, Xu C, Jin G, Chen Y, Xu X, Ma H, Chen W, Lin Y, Zheng Y, Wang J, Hu Z, Yi Y, Shen H. Clinical characteristics of 24 asymptomatic infections with COVID-19 screened among close contacts in Nanjing, China. Sci China Life Sci. 2020 May;63(5):706-711. doi: 10.1007/s11427-020-1661-4. Epub 2020 Mar 4. PMID 32146694
- [Result] Bai Y, Yao L, Wei T, Tian F, Jin DY, Chen L, Wang M. Presumed Asymptomatic Carrier Transmission of COVID-19. JAMA. 2020 Apr 14;323(14):1406-1407. doi: 10.1001/jama.2020.2565. PMID 32083643
- [Result] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501
- See also: Novel Coronavirus (2019-nCoV) situation reports — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports
- See also: World Health Organization. Coronavirus disease 2019 (COVID-19) Situation Report — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200411-sitrep-82-covid-19.pdf?sfvrsn=74a5d15_2
- See also: Guidance for discharge and ending isolation in the context of widespread community transmission of COVID-19 - first update. In: European Centre for Disease Prevention and Control — http://www.ecdc.europa.eu/en/publications-data/covid-19-guidance-discharge-and-ending-isolation